CLINICAL TRIAL: NCT04521517
Title: Addis Ababa University
Brief Title: Effect of Pamphlet Supported Counseling During Child Immunization on the Initiation of Post-partum Family Planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Dr.Sawra Getnet, Assistant professor, Family Medicine, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AddisAbabaU
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-02

CONDITIONS: Family Planning
Keywords: Postpartum; Family Planning; Intervention; Pamphlet; Ethiopia

STUDY DESIGN:
Intervention Model Description: The study will use implementation science, evaluated using a randomized control trial involving mothers coming for day 1, 6week and 10th-week vaccination of their neonate in the selected health centers, by allocating mothers randomly in two arms (the intervention and non-intervention). Mothers in the intervention arm will get thorough counseling on post-partum Family planning, will be provided with FP pamphlets in addition to the routine immunization service, while mothers from the control arms will get the routine immunization service for their babies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pamphlet with timing of family planning (Experimental): Pamphlet with timing of family planning" and "Routine service"
  Interventions: Behavioral: pamphlet describing the timing of family planning during postpartum with methods advantages and disadvantages of family planning
- Only routine service (No Intervention): Receive only routine service

INTERVENTIONS:
Behavioral: pamphlet describing the timing of family planning during postpartum with methods advantages and disadvantages of family planning — a pamphlet describing the timing of family planning during postpartum with methods advantages and disadvantages of family planning
  Arms: Pamphlet with timing of family planning

SUMMARY:
Background:- The World Health Organization (WHO) recommends postpartum family planning as a critical component of health care that has the potential to meet women's desire for contraception and save millions of maternal and infant lives in low- and middle-income countries. Family planning is known to avert a higher number of maternal deaths and child mortality. Closely spaced pregnancies within the first year postpartum are the riskiest for the mother and baby, resulting in increased risks for adverse outcomes, such as preterm, low birth weight, and small for gestational age. Adding the existing body of evidence use of intervention strategies that promote and increase postpartum family planning in the developing world is important. Therefore, this study aims to evaluate the effect of the use of pamphlet supported by counseling during child immunization in improving the overall and average time of initiation of postpartum family planning utilization in the first nine months after delivery and assess its socio-demographic predictors in selected health centers of Addis Ababa, Ethiopia Methods:- The study will use implementation science with a randomized control trial study design. The study will involve mothers coming for vaccination of their newborn child to selected three health centers that are under the catchment area of Tikur Anbessa Teaching Hospital, in Addis Ababa. Eligible mothers will be randomly assigned into intervention and non-intervention arms using computerized assignments assisted by an envelope. Mothers assigned to the interventional arm will be given a pamphlet that advises mothers about postpartum family planning followed by counseling service while women in the non-intervention arm will take the routine immunization service given in the health services. Both groups will be followed until the 9th month after the birth of the child. In the 9th month after the birth of the child, during child vaccination for measles, women will be asked for the starting date the first family planning service. A comparison of family planning service will be made between the groups using logistic regression, using bivariate and multivariable analysis. The study also will use Kaplan Meier and Cox-regression to compare the median time of postpartum family planning and its correlation using SPSS for windows version 26. The research will undertake from Dec 2019 to June 2021.

DETAILED DESCRIPTION:
Evidence shows that family planning is a cost-effective public health intervention with the potential to reduce both maternal and child mortality. However, around 222 million women have an unmet need for family planning, with the majority of these women living in low- and middle-income countries. There were 213 million pregnancies in 2012, most of which ended in birth. This number will certainly increase as the global population continues to grow, and a large proportion of youth enter their childbearing years. Regardless of whether the growing number of births are intended or unintended, they indicate an immense opportunity to reach postpartum women with family planning for spacing subsequent pregnancies. Citing the prospective definition of unmet need for family planning, which uses a postpartum woman's fertility preferences looking forward at the time of the survey, as many as 50%-90% of women from 17 low- and middle-income countries (LMICs) report an unmet need for postpartum family planning (PPFP).

Women frequently return to fertility and sex before initiating contraception after delivery and do not necessarily understand the risk of pregnancy before the return of menses. For instance, a report on Demographic and Health Survey (DHS) data showing that in Bangladesh, 33% of women resumed sexual activity within 3 months postpartum, but only 7.2% were using contraception. In Rwanda, these proportions are 73.6% and 1.7%, respectively. In all 17 countries analyzed, women were more likely to use contraception after menses returned than it was before. Therefore, family planning is critical for saving the lives of women and children in the developing world.

The World Health Organization (WHO) recommends postpartum family planning as a critical component of health care that has the potential to meet women's desire for contraception and save millions of maternal and infant lives in low- and middle-income countries.

This review aims to answer the research question: what recent interventions in LMIC have led to improvements in postpartum family planning outcomes? Therefore, the purpose of this review is to add to the existing body of evidence by casting a wide net in an attempt to capture the recent intervention strategies that present the most promise for decreasing the unmet need for contraception among postpartum women living in low- and middle-income countries (those defined as "developing" by the World Bank). The postpartum period is defined here as the 12 months after delivery. The study will assess the effectiveness of postpartum family planning (PPFP) interventions on clients' contraceptive knowledge, intention, and postpartum family planning use.

The rationale for the promotion of family planning to delay conception after a recent birth is a best practice that can lead to optimal maternal and child health outcomes. Despite the above fact uptake of postpartum family planning remains low in sub-Saharan Africa.

Therefore, the study through the use of an intervention having thorough counseling supplemented by pamphlets that will improve the awareness of women on modern use of family planning methods will improve their unmet need for family planning during postpartum time as a potential to contribute to achieving the Ethiopian Health Sector Transformation Plan and the Sustainable Development Goals. This study will help to understand the potential barriers and facilitators of PPFP uptake and the findings will be useful in modifying practice among the health care workers providing care at the maternal, neonatal, and child health (MNCH) clinics. This will create as an opportunity for the health providers and policymakers to learn to address the health needs of a community (they are working in) through a scholarly activity which is one of the family planning competencies and could be directly involved in the intervention plan to improve the gaps identified by working closer to the community.

ELIGIBILITY:
Inclusion Criteria:

* Women above the age of 18 and who are able to consent,
* Attending their child's 1st day, 6th-week or 10th-week vaccination,
* Apparently healthy, willing to continue child vaccination in the health center

Exclusion Criteria:

* Women who already started the use of contraception during the recruitment time
* Women who did permanent sterilization by hysterectomy or bilateral oophorectomy
* Women who are not the biological mother of the index child for vaccination
* Women who don't have either personal or home phone

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 346 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Family planning utilization | Time since birth to the 9th months
  Women will be assessed for utilization of modern family planning within nine months of delivering the index child [from interview and record reviewing]
The median time of family planning use | Time since birth to the 9th months
  Women will be assessed the time of initiation of family planning [from interview and record reviewing] and will be computed in weeks since the birth of the child.

REFERENCES:
- [Derived] Gelaw SG, Deyessa N, Kidane A, Evensen A, Teka A, Bokan B, Yesuf SA. Effect of postpartum family planning intervention and associated factors during child immunization in Addis Ababa, Ethiopia. Pan Afr Med J. 2024 Mar 6;47:110. doi: 10.11604/pamj.2024.47.110.34883. eCollection 2024. PMID 38766567